CLINICAL TRIAL: NCT03508102
Title: Effect of Remifentanil on the Bispectral Index in Women Undergoing Caesarean Delivery Under General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Qing Zhu, attending physician, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015001
Record Dates: First submitted 2017-11-29; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Intraoperative Awareness
Keywords: remifentanil; bispectral index; Caesarean delivery; general anesthesia
MeSH Terms: conditions — Intraoperative Awareness | interventions — Remifentanil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Remifentanil 1 μg kg-1 (R1) (Experimental): Received remifentanil 1μg/kg when induction of general anesthesia
  Interventions: Drug: remifentanil
- Remifentanil 0.5 μg kg-1 (R0.5), (Experimental): Received remifentanil 0.5μg/kg when induction of general anesthesia
  Interventions: Drug: remifentanil
- saline (control) (No Intervention): Injected the equal volume normal saline when induction of general anesthesia

INTERVENTIONS:
Drug: remifentanil — the effects of remifentanil on the average value of BIS at the time period of before induction , induction , intubation , skin incision, peritoneum incision, uterine incision, and delivery
  Other Names: saline
  Arms: Remifentanil 0.5 μg kg-1 (R0.5),; Remifentanil 1 μg kg-1 (R1)

SUMMARY:
Patients undergoing caesarean delivery under inhalation anaesthesia are at a high risk of awareness, especially in the period before delivery. The investgators assessed the effects of remifentanil on the bispectral index (BIS) in the interval before delivery.

DETAILED DESCRIPTION:
Sixty primipara undergoing elective cesarean delivery were randomly assigned to receive remifentanil 1 μg kg-1 (R1) or 0.5 μg kg-1 (R0.5), or saline (control) over 15 s with induction of anesthesia using propofol 2 mg kg-1 and suxamethonium 1.5 mg kg-1.The investgators assessed the average value of BIS at the time period of before, induction , intubation, skin incision, peritoneum incision , uterine incision , and delivery. The investgators also determined the neonatal Apgar scores, and conducted umbilical artery blood gas analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II who elected to undergo Caesarean section, under general anaesthesia

Exclusion Criteria:

* multiple fetuses,preterm delivery, known fetal anomalies, pregnancy-induced hypertension, or any other medical complication

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
the effects of remifentanil on the bispectral index (BIS) in the interval before delivery. | the time of before induction, induction , intubation, skin incision, peritoneum incision , uterine incision , and delivery
  the average value of BIS at the time period of before induction, induction , intubation, skin incision, peritoneum incision , uterine incision , and delivery

SECONDARY OUTCOMES:
incidence of intraoperative awareness | one day and one week after delivery.
  the maternal incidence of intraoperative awareness